CLINICAL TRIAL: NCT03115736
Title: Prospective Cohort Study to Assess the Safety and Efficacy of Replacing Tenofovir Disoproxil Fumarate by Tenofovir Alafenamide in HIV/HBV-coinfected Patients With Mild or Moderate Renal Dysfunction
Brief Title: TAF for HIV-HBV With Renal Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSEL-HINF-2017-1
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: HIV and Hepatitis B Coinfection
Keywords: HIV; Hepatitis B; Renal dysfunction; tenofovir alafenamide
MeSH Terms: conditions — Hepatitis B; Renal Insufficiency | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Switch (Experimental): Patients are switched from a TDF-containing antiretroviral therapy regimen to a TAF-containing regimen
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Patients are switched to either Genvoya (TAF/FTC/EVG/COB) or another FTC/TAF-containing ART regimen

SUMMARY:
The investigators aim at describing changes in renal glomerular and tubular function with after the switch from TDF to TAF in HIV/HBV-coinfected patients with mild to moderate renal dysfunction and to assess the virological efficacy of TAF on HBV infection.

The study will include HIV/HBV-coinfected participants of the Swiss HIV Cohort Study (SHCS) who are under active care and have been on a stable, TDF-containing ART regimen for at least 6 months. Only patients with an estimated glomerular filtration rate (GFR) between 30 ml/min and 90 ml/min will be included. All individuals who agree to participate will be switched from a TDF-containing ART regimen to a TAF-containing triple ART regimen at week 0 and will be followed for 48 weeks after the treatment change.

DETAILED DESCRIPTION:
Rationale:

Tenofovir alafenamide (TAF) has been shown to cause less renal complications than tenofovir disoproxil fumarate (TDF) while having the same virological efficacy against HIV and HBV infections. In a recent study from the USA and Japan, over 90% of HIV/HBV-coinfected individuals had a suppressed HBV viral load 48 weeks after TDF was replaced by TAF. Thus, TAF might be a valuable treatment option for HIV/HBV-coinfected individuals with TDF-toxicity, especially in the context of resistance to lamivudine and entecavir. However, the safety and efficacy of TAF has not been evaluated to date in HIV/HBV-coinfected patients with renal dysfunction.

Primary objectives:

* To evaluate changes in glomerular and tubular renal function after switch from TDF to TAF in HIV/HBV coinfected patients with renal dysfunction
* To assess the HBV virological efficacy of TAF in HIV/HBV coinfected patients with renal dysfunction switching from TDF to TAF.

Secondary objectives:

* To assess the percentage of and reasons for treatment interruptions
* To describe toxicity events including liver-related complications
* To evaluate changes in liver fibrosis

Intervention:

In eligible patients willing to participate and who have signed an informed consent TDF will be replaced by TAF on day 1 of the study.

Products:

* Tenofovir alafenamide/emtricitabine (TAF/FTC) Dose: one tbl. once per day in addition to at least one third compound OR
* Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (EVG/COBI/FTC/TAF) Dose: one tbl. once per day

Study Population: eligible patients from all 7 centers of the Swiss HIV Cohort Study will be considered.

ELIGIBILITY:
Inclusion Criteria:

* HIV/HBV-coinfection
* Suppressed HIV-viremia (<200 cp/ml)
* On TDF-containing ART since at least 6 months
* eGFR > 30 ml/min and <90 ml/min
* Written informed consent

Exclusion Criteria:

* Study drug considered by the treating physician not a valid option for the patient
* Pregnancy
* Decompensated liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change in renal function | 48 weeks
  Assessment of change in eGFR and tubular markers during the first year of TAF-containing ART
HBV suppression | 48 weeks
  Evaluation of HBV virological suppression and HBsAg loss after 12 months of TAF

SECONDARY OUTCOMES:
Treatment interruptions | 48 weeks
  Description of the proportion of patients with treatment changes or interruptions
Adverse events | 48 weeks
  Evaluation of the proportion of patients with adverse events during therapy, including grade 2 or above transaminases elevations
Liver fibrosis change | 48 weeks
  Assessment of the proportion of patients with a change in liver fibrosis stage

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Wandeler, MD MSc, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (8):
- Switzerland (8):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Cabinet médical Chave-Crottaz-Roggerto, Lausanne, Canton of Vaud
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne, Vaude
  - Klinik für Infektiologie und Spitalhygiene, Universitätspital Basel, Basel
  - Inselspital, Bern
  - Department of Infectious Diseases, Hôpitaux Universitaires de Genève, Geneva
  - Klinik für Infektionskrankheiten & Spitalhygiene, Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Surial B, Beguelin C, Chave JP, Stockle M, Boillat-Blanco N, Doco-Lecompte T, Bernasconi E, Fehr J, Gunthard HF, Schmid P, Walti LN, Furrer H, Rauch A, Wandeler G; and the Swiss HIV Cohort Study. Brief Report: Switching From TDF to TAF in HIV/HBV-Coinfected Individuals With Renal Dysfunction-A Prospective Cohort Study. J Acquir Immune Defic Syndr. 2020 Oct 1;85(2):227-232. doi: 10.1097/QAI.0000000000002429. PMID 32925387